CLINICAL TRIAL: NCT02205879
Title: Double Blind Placebo Controlled Randomized Clinical Trial of Pregabalin for Alcohol Dependence
Brief Title: Pregabalin for Alcohol Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Petersburg Bekhterev Research Psychoneurological Institute (Other)
Collaborators: St.-Petersburg Bekhterev Research Psychoneurological Institute, Russian Federation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BRPI-PGBL-A01
Record Dates: First submitted 2014-07-30; First posted 2014-07-31 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Alcoholism
Keywords: pregabalin; patients; treatment
MeSH Terms: conditions — Alcoholism | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pregabalin (Experimental)
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin
  Arms: pregabalin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study hypothesis is: Pregabalin is superior to placebo in preventing relapse to drinking and reducing drinking severity

DETAILED DESCRIPTION:
This is a two cell double blind placebo controlled randomized clinical trial of pregabalin for alcohol dependence

ELIGIBILITY:
Inclusion Criteria:

* Alcohol Dependence by ICD-X criteria

Exclusion Criteria:

* Severe co-morbid psychiatric and somatic diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Retention in treatment | three months
  Number of subjects retianed in treatment (not relapsed)

SECONDARY OUTCOMES:
Weekly alcohol consumption | three months
  Time Line Follow Back technique

OTHER OUTCOMES:
Anxiety | three months
  Hamilton anxiety scale and Spielbereger State Trait Anxiety test

CONTACTS AND LOCATIONS:
Locations (1):
- St.-Petersburg Bekhterev Reserach Psychoneurological Institute, Saint Petersburg, Russia